CLINICAL TRIAL: NCT01846169
Title: Healthy Eating for At-Risk Older Adults (HERO)
Brief Title: Study to Improve Healthy Eating for At-Risk Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUN-12-2011-004
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Biometrics
Keywords: food insecurity; older adults; nutrition; food deliveries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- food deliveries (Experimental): After baseline screening, participants receive weekly or bi-weekly food deliveries and brief nutrition education.
  Interventions: Behavioral: Food deliveries

INTERVENTIONS:
Behavioral: Food deliveries — Frequency of food deliveries is based on level of food insecurity at baseline (i.e., more food insecurity receives more frequent food deliveries). Deliveries are tailored to the diet of the client (e.g., consist of soft foods if participant has trouble chewing; has more fruits and vegetables if that was a food category the participant at less of at baseline). The brief nutrition education is a review of basic nutrition concepts and healthy eating ideas.

SUMMARY:
This application, funded by the American Association of Retired Persons(AARP) Foundation, is to implement the Healthy Eating for at Risk Older Adults (HERO) initiative. This initiative will address barriers of affordability, and reduced mobility by providing older adults with nutritious foods that are usually difficult to purchase due to high cost; delivering needed foods to individuals in their homes; tailoring food delivery frequency based on level of food insecurity; and offering basic nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older
* if member of Boston Medical Center's Elders Living at Home Program: Not currently homeless and expect to live at current residence or in the area for next 6 months
* if NOT member of Boston Medical Center's Elders Living at Home Program: Not currently homeless, live at public housing development, and plan to live there for at least next 6 months
* Able to understand, speak and read English

Exclusion Criteria:

* Follows a special diet that cannot be accommodated, as ascertained by clinical judgment of the nurse.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
body composition | 6 months
  percent body fat
BMI | 6 months
  Body mass index
weight | 6 months
  total body weight in pounds
blood pressure | 6 months
  systolic and diastolic blood pressure
blood glucose | 6 months
  measurement of blood glucose

SECONDARY OUTCOMES:
nutritional risk | 6 months
  food frequency questionnaire assessing levels of food intake in pre-specified categories (e.g., fruits and vegetables)
food insecurity | 6 months
  measurement of food insecurity as assessed by standard questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Brien, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: AARP Foundation — http://www.aarp.org/aarp-foundation/